CLINICAL TRIAL: NCT02512016
Title: Bridging Physical and Cultural Determinants of Postpartum Pelvic Floor Support and Symptoms Following Vaginal Delivery
Brief Title: Motherhood and Pelvic Health (MAP Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ingrid Nygaard, M.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 82389
Record Dates: First submitted 2015-07-16; First posted 2015-07-30 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Postpartum Pelvic Floor Function and Symptoms
Keywords: Pelvic floor
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nulliparous Women in Third Trimester (Other): Study Procedures
  Interventions: Other: Study Procedures

INTERVENTIONS:
Other: Study Procedures — * Pelvic Organ Prolapse Quantification exam (3rd tri, 8 wks and 1 yr postpartum)
  * Intra-abdominal pressure measure. At 8 weeks: IAP during lifting 12.5 kg and abdominal muscle endurance testing. At 1 year: IAP during lifting 17.5 kg and abdominal muscle endurance testing.
  * Accelerometry: Wrist accelerometer (objective quantification of physical activity) x 1 wk 2-3 and 5-6 wks and 6 mo postpartum.
  * Measures of strength and body habitus:
    8 weeks and 1 year postpartum: Abdominal muscle endurance Abdominal adiposity Body mass index
    1 year postpartum: Pelvic floor muscle strength: tested using a Peritron manometer Body composition: using air displacement plethysmography using the BodPod
  * Qualitative interviews: A smaller number of participants will be purposefully selected for the qualitative interviews in order to understand examples of the postpartum sensations and experiences of women with a wide variety of characteristics and from various social and cultural settings.

SUMMARY:
The Motherhood and Pelvic health study (MAP), Bridging physical and cultural determinants of postpartum pelvic floor support and symptoms following vaginal delivery, uses mixed methods research to study the influences of intra-abdominal pressure, physical activity and strength on pelvic floor support and symptoms and the cultural context in which women experience those changes.

DETAILED DESCRIPTION:
Vaginal delivery affects pelvic muscles, nerves and connective tissue. Despite the similarities between vaginal delivery and other non-pelvic soft tissue injuries, research to date has not focused on factors related to recovery from childbirth, but instead has been directed at intrapartum interventions. A woman's pelvic floor derives its ability to withstand loads from physical activities due to her inherent genetic make-up that sets the foundation for her muscle, connective tissue, bone and other structures, her history of injury, and her ability to recover from injuries. Over the past decade, investigators have gained important information about some of the ways in which vaginal delivery affects the structure and function of the pelvic floor.

However, investigators know very little about how pelvic floor function recovers after vaginal delivery. This study will look at whether the non-pregnant milieu, including physical and cultural factors, mediate the effects of vaginal childbirth. Study investigators propose that pelvic floor support and symptoms 1 year after the first vaginal delivery are affected by biologically plausible factors that may impact muscle, nerve and connective tissue healing during the postpartum recovery period (first 8 weeks postpartum) and pelvic floor function during the postpartum strengthening period (remainder of the first postpartum year): in particular, timing and dose of moderate/vigorous physical activity and inactivity, and timing of and exposure to a range of intra-abdominal pressures. Our investigators further propose that perception of pelvic floor support and symptoms 1 year after vaginal delivery are influenced by cultural attributes and beliefs. Finding relationships between physical activity, muscular strength, intra-abdominal pressure and pelvic floor support /symptoms will provide realistic targets for disease prevention and pelvic floor health management.

Hispanics are the fastest-growing ethnic group in the United States. Although the risks for pelvic floor disorders differ among ethnic and racial groups, few studies have examined these differences. There is a critical need for research among Hispanic women. In this Program, our investigators will study personal and cultural aspects of Mexican-American and Euro-American primiparas' experiences of the earliest changes that happen after childbirth and make them understandable to women and clinicians, creating an opportunity for dialogue across lay and medical discourses.

The aims of each project are summarized below.

PROJECT 1 Intra-abdominal pressure and postpartum pelvic floor support and symptoms

By using an intra-vaginal sensor to measure intra-abdominal pressure in primiparous women, investigators will:

Aim 1: Determine whether IAP measured at 8 weeks postpartum during a) lifting and b) abdominal muscle endurance testing predicts pelvic floor support and symptoms 1 year postpartum.

Aim 2: Determine whether measures of muscular fitness modify the effect of IAP during lifting on pelvic floor support at 1 year postpartum.

PROJECT 2: Physical activity, inactivity, and fitness: Impact on postpartum pelvic floor support and symptoms

Aims: To determine, in primiparous women after vaginal delivery, whether physical activity, sedentary time and the characteristics of body habitus and muscular fitness are associated with 1) pelvic floor support and 2) pelvic floor symptoms 1 year postpartum.

PROJECT 3: The cultural context of postpartum pelvic floor support following vaginal delivery: a comparative ethnographic analysis of Mexican-American and Euro-American women.

Aim: To describe primiparous Mexican-American and Euro-American women's experiences and cultural knowledge of postpartum pelvic floor support changes.

Sub-aim 1: To characterize the ways women perceive and make sense of early changes in pelvic floor support as well as the ways they use language and discourse to construct meaning about those changes in the year after their first delivery.

Aim 1.2: To describe how primipara share experiences and cultural understandings of postpartum pelvic floor support with mothers, partners, sisters, and confidantes in their families and social networks.

Sub-aim 1: To explore the interplay of women's understandings of early changes in pelvic floor support with sociocultural prescriptions/proscriptions regarding physical activity and any resulting postpartum alterations of activity which they may undertake.

Estimated enrollment: 1530 women in third trimester to obtain final enrollment goal of 585 women at 1 year postpartum. (We estimate that, after initial enrollment, we will exclude 26.5% that deliver by cesarean, 10% that deliver before 37 weeks, and that 20% will withdraw between delivery and 8 weeks postpartum, 20% will withdraw between 8 weeks and 1 year postpartum, and 6% will have known pregnancy by 1 year postpartum, leaving 585 with final 1-year data.)

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Estimated gestational age 28 weeks to 36 6/7 weeks
* Nulliparous
* Single gestation

Exclusion Criteria:

* Obstructive pulmonary disease
* Collagen disorder such as Marfan's or Ehlers-Danlos
* Muscular dystrophy
* Prior surgical procedure for urinary incontinence or pelvic organ prolapse
* Required ambulatory aid before pregnancy
* No access to telephone or computer during course of study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1079 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Support | 1 Year postpartum
  Assessed using the Pelvic Organ Prolapse Quantification examination, categorized into maximum vaginal descent at or below the hymen (>/= 0 cm) versus above the hymen (< 0 cm)
Pelvic Floor symptoms | 1 Year postpartum
  Assessed using the Epidemiology of Prolapse and Incontinence Questionnaire, dichotomized as the presence of symptoms accompanied by at least minimal bother (>0 on the visual analogue scale) in at least 2 (vs 0 or 1) of the 6 domains

SECONDARY OUTCOMES:
Symptoms of Stress Urinary Incontinence | 1 Year
  Symptom of stress urinary incontinence at 1 year, assessed using the Epidemiology of Prolapse and Incontinence Questionnaire
Urinary Incontinence Severity | 1 Year
  Urinary incontinence severity at 1 year, assessed using the Incontinence Severity Index
Overactive Bladder Symptoms | 1 Year
  Symptom of overactive bladder at 1 year, assessed using the Epidemiology of Prolapse and Incontinence Questionnaire
Constipation Symptoms | 1 Year
  Constipation at 1 year, assessed using the Defecation Distress Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Nygaard, MD, Study Director — University of Utah; Marlen Egger, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Ryan JT, Day H, Egger MJ, Wu J, Depner CM, Shaw JM. Night-time sleep duration and postpartum weight retention in primiparous women. Sleep Adv. 2023 Dec 27;5(1):zpad056. doi: 10.1093/sleepadvances/zpad056. eCollection 2024. PMID 38314118